CLINICAL TRIAL: NCT01448044
Title: A Phase 3 Evaluation of BMS-790052 in Combination With Peg-Interferon Alfa-2a and Ribavirin in Treatment Naive Subjects With Chronic Hepatitis C Genotype 4
Brief Title: Phase III BMS-790052 Add-On to Peg-Interferon Alfa-2a and Ribavirin in Naive Hepatitis C
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AI444-042; 2011-002793-23 (EudraCT Number)
Record Dates: First submitted 2011-10-05; First posted 2011-10-07 (Estimated); Results first posted 2015-09-07 (Estimated); Last update posted 2015-10-12 (Estimated); Status verified 2015-09

CONDITIONS: Hepatitis C
Keywords: hepatitis C virus
MeSH Terms: conditions — Hepatitis C | interventions — daclatasvir; peginterferon alfa-2a; Ribavirin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- BMS-790052 + PegIFNα-2a + Ribavirin (Experimental): * BMS-790052 60 mg Tablets, Oral, once daily for 24 weeks
  * PegIFNα-2a 180 μg Subcutaneous Injection, once weekly for 24 or 48 weeks depending on response
  * Ribavirin 400 mg (2 tablets for participants < 75 kg) or 600 mg (3 tablets for participants ≥ 75 kg) in the morning and 600 mg (3 tablets) in the evening, Oral for 24 or 48 weeks depending on response
  Interventions: Drug: BMS-790052 (NS5A Replication Complex Inhibitor); Drug: Pegylated-interferon alfa 2a; Drug: Ribavirin
- Placebo matching BMS-790052 + PegIFNα-2a + Ribavirin (Placebo Comparator): * Placebo matching BMS-790052 0 mg Tablets, Oral, once daily for 48 weeks
  * PegIFNα-2a 180 μg Subcutaneous Injection, once weekly for 48 weeks
  * Ribavirin 400 mg (2 tablets for participants < 75 kg) or 600 mg (3 tablets for participants ≥ 75 kg) in the morning and 600 mg (3 tablets) in the evening, Oral for 48 weeks
  Interventions: Drug: Placebo matching BMS-790052; Drug: Pegylated-interferon alfa 2a; Drug: Ribavirin

INTERVENTIONS:
Drug: BMS-790052 (NS5A Replication Complex Inhibitor)
  Arms: BMS-790052 + PegIFNα-2a + Ribavirin
Drug: Placebo matching BMS-790052
  Arms: Placebo matching BMS-790052 + PegIFNα-2a + Ribavirin
Drug: Pegylated-interferon alfa 2a
  Other Names: Pegasys
Drug: Ribavirin
  Other Names: Copegus

SUMMARY:
The purpose of this study is to compare the sustained virologic response at post treatment Week 12 for each cohort (BMS-790052/Pegylated-interferon alfa 2a (pegIFNα-2a)/Ribavirin (RBV) versus placebo/PegIFNα-2a/RBV).

ELIGIBILITY:
Inclusion Criteria:

* Participants chronically infected with HCV Genotype 4
* HCV RNA viral load of ≥ 10,000 IU/mL
* No previous exposure to an interferon formulation, RBV or HCV direct antiviral agent
* Results of a liver biopsy obtained within three years prior to enrollment to demonstrate the absence of cirrhosis. Participants with compensated cirrhosis are permitted, however, and any prior biopsy is permitted

Exclusion Criteria:

* Evidence of decompensated liver disease
* Documented or suspected Hepatocellular carcinoma (HCC)
* Positive for Hepatitis B surface antigen (HBsAg) or Human immunodeficiency virus-1 (HIV-1)/HIV-2 antibody at screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2011-12; Primary Completion 2013-10 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (22):
- United States (4):
  - Scti Research Foundation, San Clemente, California
  - Umass Memorial Medical Center, Worcester, Massachusetts
  - University Gastroenterology, Providence, Rhode Island
  - Metropolitan Research, Annandale, Virginia
- France (10):
  - Local Institution, Bondy
  - Local Institution, Créteil
  - Local Institution, La Roche-sur-Yon
  - Local Institution, Marseille
  - Local Institution, Nice
  - Local Institution, Orléans
  - Local Institution, Paris
  - Local Institution, Strasbourg
  - Local Institution, Toulouse
  - Local Institution, Villejuif
- Local Institution, Thesaloniki, Greece
- Italy (2):
  - Local Institution, Roma
  - Local Institution, Torino
- Local Institution, San Juan, Puerto Rico
- Spain (3):
  - Local Institution, A Coruña
  - Local Institution, Barcelona
  - Local Institution, Madrid
- Local Institution, London, Greater London, United Kingdom

REFERENCES:
- [Derived] Hezode C, Alric L, Brown A, Hassanein T, Rizzetto M, Buti M, Bourliere M, Thabut D, Molina E, Rustgi V, Samuel D, McPhee F, Liu Z, Yin PD, Hughes E, Treitel M; COMMAND-4 study team. Randomized controlled trial of the NS5A inhibitor daclatasvir plus pegylated interferon and ribavirin for HCV genotype-4 (COMMAND-4). Antivir Ther. 2015 Aug 27;21(3):195-205. doi: 10.3851/IMP2985. Online ahead of print. PMID 26313445
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 152 participants were enrolled in the study, of which 125 were randomized and 27 participants were not randomized due to 23 no longer met criteria, 1 withdrew consent, 1 due to administrative reason, and 2 other reasons. Of 125 randomized, 124 were treated and 1 was not treated due to withdrawal of consent.
Groups:
- Daclatasvir + PegIFNα2a + Ribavirin: Daclatasvir 60 mg tablets were administered orally once daily for 24 weeks, peginterferon alfa-2a (PegIFNα2a) 180 µg was administered subcutaneously once in a week for 24 or 48 weeks depending on response and ribavirin 400 mg (2 tablets for participants <75 kg) or 600 mg (3 tablets for participants >=75 kg) was administered orally in the morning and 600 mg (3 tablets) in the evening for 24 or 48 weeks depending on response.
- Placebo + PegIFNα2a + Ribavirin: Placebo matching daclatasvir tablets was administered orally once daily for 48 weeks. Peginterferon alfa-2a (PegIFNα2a) 180 µg was administered subcutaneously once in a week for 48 weeks and ribavirin 400 mg (2 tablets for participants <75 kg) or 600 mg (3 tablets for participants >=75 kg) was administered orally in the morning and 600 mg (3 tablets) in the evening for 48 weeks.
Period: Treatment Period
Arm/Group | Daclatasvir + PegIFNα2a + Ribavirin | Placebo + PegIFNα2a + Ribavirin
Started | 82 | 42
Completed | 59 | 26
Not Completed | 23 | 16
Not completed — Adverse Event | 4 | 3
Not completed — Lack of Efficacy | 5 | 12
Not completed — Subject requested discontinue study drug | 1 | 0
Not completed — Completed 24 weeks treatment period only | 8 | 0
Not completed — Participant does not meet study criteria | 1 | 0
Not completed — Lost to Follow-up | 2 | 1
Not completed — Other reason | 2 | 0
Period: Follow Up Period
Arm/Group | Daclatasvir + PegIFNα2a + Ribavirin | Placebo + PegIFNα2a + Ribavirin
Started | 77 (Out of 82 participants who entered the treatment period, 77 continued in the follow-up period.) | 40 (Out of 42 participants who entered the treatment period, 40 continued in the follow-up period.)
Completed | 65 | 26
Not Completed | 12 | 14
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Lost to Follow-up | 6 | 2
Not completed — Other | 5 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Daclatasvir + PegIFNα2a + Ribavirin | Placebo + PegIFNα2a + Ribavirin | Total
Number analyzed (Participants) | 82 | 42 | 124
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.7 (10.23) | 48.4 (8.09) | 48.0 (9.53)
Age, Customized [Number; unit: participants]
  < 21 years | 1 | 0 | 1
  21 to < 65 years | 78 | 42 | 120
  >= 65 years | 3 | 0 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 13 | 34
  Male | 61 | 29 | 90

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With 12 Week Sustained Virologic Response (SVR12)
Description: Participants were assessed for sustained virologic response 12 weeks post treatment (SVR12) defined as hepatitis C virus (HCV) RNA levels < lower limit of quantitation (LLOQ was 25 IU/mL), target detected (TD) or target not detected (TND) at post-treatment Week 12.
Time Frame: Week 12 (Follow-up period)
Population: The analysis was performed in modified Intent to treat population (ITT), defined as the proportions of participants meeting the response criteria in numerator and denominator based on all treated participants. Missing values were imputed using backward imputation technique.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Daclatasvir + PegIFNα2a + Ribavirin | Placebo + PegIFNα2a + Ribavirin
Number analyzed (Participants) | 82 | 42
Percentage of participants | 81.7 [73.3 to 90.1] | 42.9 [27.9 to 57.8]
Statistical Analysis 1: Comparison: Daclatasvir + PegIFNα2a + Ribavirin vs Placebo + PegIFNα2a + Ribavirin; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — The pvalue was based on the CochranMantelHaenszel (CMH) test, stratified by IL28B host genotype, geography, and baseline cirrhosis status; difference in percentages = 38.850, 95% CI 2-sided [21.703 to 55.997]

2. Secondary Outcome: Percentage of Participants Who Achieve HCV Ribonucleic Acid (RNA) < Limit of Quantification (LLOQ)
Description: Participants who achieved HCV RNA levels below LLOQ ie, 25 international unit per milliliter (IU/mL). Participants in the placebo arm did not have visits beyond post treatment Week 24.
Time Frame: Treatment Weeks 1, 2, 4, 6, 8 and 12; Weeks 4 and 12; End of treatment (EOT); Post treatment Week 24; Post treatment Week 48
Population: The analysis was performed in modified ITT population.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Daclatasvir + PegIFNα2a + Ribavirin | Placebo + PegIFNα2a + Ribavirin
Number analyzed (Participants) | 82 | 42
Percentage of participants
  Week 1 | 53.7 [42.9 to 64.5] | 4.8 [0.0 to 11.2]
  Week 2 | 89.0 [82.3 to 95.8] | 11.9 [2.1 to 21.7]
  Week 4 | 91.5 [85.4 to 97.5] | 19.0 [7.2 to 30.9]
  Week 6 | 84.1 [76.2 to 92.1] | 40.5 [25.6 to 55.3]
  Week 8 | 87.8 [80.7 to 94.9] | 47.6 [32.5 to 62.7]
  Week 12 | 85.4 [77.7 to 93.0] | 59.5 [44.7 to 74.4]
  Weeks 4 and 12 | 84.1 [76.2 to 92.1] | 19.0 [7.2 to 30.9]
  End of Treatment | 92.7 [87.0 to 98.3] | 64.3 [49.8 to 78.8]
  Post treatment Week 24 | 80.5 [71.9 to 89.1] | 40.5 [25.6 to 55.3]
  Post treatment Week 48 | 83.6 [73.9 to 93.4] | NA [NA to NA] — No visit on post treatment Week 48 was planned for this arm.

3. Secondary Outcome: Percentage of Participants With Undetectable Hepatitis C Virus (HCV) RNA Levels
Description: Participants who achieved HCV RNA undetectable ie, 10 international units per milliliter (IU/mL). Participants in the placebo arm did not have visits beyond post treatment Week 24.
Time Frame: Treatment Weeks 1, 2, 4, 6, 8 and 12; Weeks 4 and 12, End of treatment (EOT), Post treatment Week 24, Post treatment Week 48
Population: The analysis was performed in modified ITT population.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Daclatasvir + PegIFNα2a + Ribavirin | Placebo + PegIFNα2a + Ribavirin
Number analyzed (Participants) | 82 | 42
Percentage of participants
  Week 1 | 14.6 [7.0 to 22.3] | 0.0 [0.0 to 0.0]
  Week 2 | 45.1 [34.4 to 55.9] | 9.5 [0.6 to 18.4]
  Week 4 | 85.4 [77.7 to 93.0] | 11.9 [2.1 to 21.7]
  Week 6 | 80.5 [71.9 to 89.1] | 16.7 [5.4 to 27.9]
  Week 8 | 87.8 [80.7 to 94.9] | 38.1 [23.4 to 52.8]
  Week 12 | 84.1 [76.2 to 92.1] | 47.6 [32.5 to 62.7]
  Weeks 4 and 12 (VR 4 & 12) | 79.3 [70.5 to 88.0] | 11.9 [2.1 to 21.7]
  EOT | 90.2 [83.8 to 96.7] | 64.3 [49.8 to 78.8]
  Post treatment Week 24 | 78.0 [69.1 to 87.0] | 40.5 [25.6 to 55.3]
  Post treatment Week 48 | 81.8 [71.6 to 92.0] | NA [NA to NA] — No visits planned for post treatment Week 48 for this arm.

4. Secondary Outcome: Percentage of Participants With Sustained Virologic Response at Follow-up Week 12 (SVR12) or Sustained Virologic Response at Follow-up Week 24 (SVR24) by rs12979860 Single Nucleotide Polymorphism (SNP) in the IL28B Gene
Description: Participants categorized into three genotypes based on SNPs in the IL28B gene were assessed for SVR12 and SVR24, defined as response in which hepatitis C virus RNA levels below lower limit of quantitation or below target detected or target not detected at follow-up Week 12 and Week 24 respectively.
Time Frame: Post Treatment Weeks 12, 24
Population: For SVR12; analysis was performed by backward imputation method, For SVR24: analysis was performed in Modified ITT population.
Measure: Number; unit: Percentage of participants
Arm/Group | Daclatasvir + PegIFNα2a + Ribavirin | Placebo + PegIFNα2a + Ribavirin
Number analyzed (Participants) | 82 | 42
Percentage of participants
  IL28B Genotype CC (SVR12) (n=22, 9) | 95.5 | 100.0
  IL28B Genotype CT (SVR12) (n=40, 27) | 75.0 | 33.3
  IL28B Genotype TT (SVR12) (n=20, 6) | 80.0 | 0.0
  IL28B Genotype CC (SVR24) (n=22, 9) | 95.5 | 88.9
  IL28B Genotype CT (SVR24) (n=40, 27) | 72.5 | 33.3
  IL28B Genotype TT (SVR24) (n=20, 6) | 80.0 | 0.0

5. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs), Discontinuations Due to Adverse Events (AEs) and Who Died
Description: AE was defined as any new unfavorable symptom, sign, or disease or worsening of a pre-existing condition that does not necessarily have a causal relationship with treatment. SAE was defined as a medical event that at any dose resulted in death, persistent or significant disability/incapacity, was life-threatening, an important medical event, or a congenital anomaly/birth defect; or required or prolonged hospitalisation.
Time Frame: From Day 1 (start of study treatment) up to Follow-up Week 4
Population: Analysis was performed on all treated participants.
Measure: Number; unit: participants
Arm/Group | Daclatasvir + PegIFNα2a + Ribavirin | Placebo + PegIFNα2a + Ribavirin
Number analyzed (Participants) | 82 | 42
participants
  AEs leading to discontinuation of study drug | 4 | 3
  SAEs | 8 | 2
  Death | 0 | 0

ADVERSE EVENTS:
Time Frame: From first dose to last dose plus 7 days (baseline up to 49 weeks)
Description: on-treatment
Arm/Group | Daclatasvir + PegIFNα2a + Ribavirin | Placebo + PegIFNα2a + Ribavirin
Serious Adverse Events (participants affected / at risk) | 8/82 | 2/42
Other Adverse Events (participants affected / at risk) | 80/82 | 39/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Daclatasvir + PegIFNα2a + Ribavirin (N=82) | Placebo + PegIFNα2a + Ribavirin (N=42)
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 2 | 0
Basedow's disease (Endocrine disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 | 0
Thyroid cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bile duct stone (Hepatobiliary disorders) | 0 | 1
Cluster headache (Nervous system disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Daclatasvir + PegIFNα2a + Ribavirin (N=82) | Placebo + PegIFNα2a + Ribavirin (N=42)
Dry skin (Skin and subcutaneous tissue disorders) | 12 | 7
Eczema (Skin and subcutaneous tissue disorders) | 3 | 4
Abdominal pain upper (Gastrointestinal disorders) | 7 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 10 | 8
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 8
Rash (Skin and subcutaneous tissue disorders) | 15 | 8
Anaemia (Blood and lymphatic system disorders) | 20 | 12
Dry mouth (Gastrointestinal disorders) | 3 | 3
Erythema (Skin and subcutaneous tissue disorders) | 2 | 5
Influenza like illness (General disorders) | 23 | 13
Myalgia (Musculoskeletal and connective tissue disorders) | 15 | 11
Decreased appetite (Metabolism and nutrition disorders) | 20 | 5
Diarrhoea (Gastrointestinal disorders) | 7 | 4
Irritability (General disorders) | 11 | 9
Pruritus (Skin and subcutaneous tissue disorders) | 25 | 13
Dry eye (Eye disorders) | 3 | 4
Dyspepsia (Gastrointestinal disorders) | 3 | 3
Neutropenia (Blood and lymphatic system disorders) | 12 | 11
Pyrexia (General disorders) | 13 | 8
Anxiety (Psychiatric disorders) | 3 | 4
Asthenia (General disorders) | 47 | 25
Back pain (Musculoskeletal and connective tissue disorders) | 11 | 6
Constipation (Gastrointestinal disorders) | 2 | 3
Fatigue (General disorders) | 6 | 7
Insomnia (Psychiatric disorders) | 18 | 6
Nausea (Gastrointestinal disorders) | 10 | 5
Abnormal loss of weight (Metabolism and nutrition disorders) | 5 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 | 6
Alopecia (Skin and subcutaneous tissue disorders) | 7 | 2
Depression (Psychiatric disorders) | 3 | 3
Headache (Nervous system disorders) | 28 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.